CLINICAL TRIAL: NCT05396872
Title: A Multi-stage Study to Improve Informed Decision-making for Precision Oncology in Veterans With Advanced Prostate Cancer
Brief Title: Patient Decision-making About Precision Oncology in Veterans With Advanced Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22554; NCI-2022-04352 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Advanced Prostate Carcinoma
Keywords: Informed Decision-Making; Precision Oncology; Military Veterans; Germline Testing; Somatic Testing; Targeted Therapy; Genetic Testing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLOSED TO ENROLLMENT: Stage 1 & 2: Patients, Caregivers, Providers (Experimental): Patient participants will be instructed to install a mobile app to record their medical appointment, which research staff will use to analyze patient-provider communication. All participants will undergo semi-structured interviews and/or focus groups. Post appointment follow-up with surveys and assessments regarding knowledge of disease information, quality of life, and other measures will be administered after the provider-patient appointment.
  Interventions: Other: Participant Surveys; Other: Mobile app
- Stage 3: Patients, Caregivers using developed GA platform (Experimental): About 14 days prior to scheduled germline testing appointment, patients and caregivers call or meet with a coach to select decision aid GA platform preference delivery (online, print, or both online and print), review the GA online platform, and possibly undergo consultation and training for audio recording of the scheduled appointment. Patients and caregivers attend the scheduled germline testing appointment on day 1. Patients complete surveys and patients and caregivers may complete an interview on study. Providers participate in focus groups and complete surveys on study.
  Interventions: Other: Participant Surveys; Other: Mobile app

INTERVENTIONS:
Other: Participant Surveys — Online surveys administered post appointment
Other: Mobile app — Mobile application installed on mobile device

SUMMARY:
This clinical trial explores and implements methods to improve informed decision making (IDM) regarding precision oncology tests amongst veterans with prostate cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Precision oncology, the use of germline genetic testing and tumor-based molecular assays to inform cancer care, has become an important aspect of evidence-based care for men with advanced prostate cancer. Veterans with metastatic castrate-resistant prostate cancer may not be carrying out IDM due to unmet decisional needs. An informed decision is a choice based on complete and accurate information. The information gained from this study will help researchers develop a decision support intervention (DSI) and implement the intervention. A DSI may serve as a valuable tool to reduce ongoing racial disparities in genetic testing and encourage enrollment to precision oncology trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate patient-participants' decisional conflict about precision oncology. (Stage I)

II. To develop a Decision Support Intervention (DSI) to improve decision-making about precision oncology. (Stage II)

III. To evaluate the percentage of invited participants who enroll. (Stage III)

SECONDARY OBJECTIVES:

I. To evaluate patient-participants' precision oncology knowledge. (Stage I).

II. To evaluate patient-participants' perceived shared decision-making effort. (Stage I)

III. To evaluate the degree of decision support provided by provider-participants during an appointment with the patient-participant. (Stage I)

IV. To evaluate patient-participants' and caregiver-participants' decisional needs, potential solutions, and potential disparities about precision oncology. (Stage I)

V. To evaluate patient-participants' decisional needs, and to identify potential disparities about precision oncology from the perspective of the provider-participant. (Stage I)

VI. To evaluate how many patient-participants receive a precision oncology intervention or testing after having an appointment and discussion with a provider-participant. (Stage I)

VII. To describe the multi-stakeholder development process of the DSI. (Stage II)

VIII. To evaluate change in participant informed decision-making about germline testing after provision of a decision support intervention. (Stage III)

IX. To evaluate the percent of intervention agents (people who deliver the intervention) who are willing to initiate the decision support intervention. (Stage III)

X. To evaluate intervention agents' (people who deliver the intervention) fidelity to the various elements of the decision support intervention. (Stage III)

XI. To evaluate patient-participant uptake of the decision support intervention. (Stage III)

XII. To measure patient-participant satisfaction with the decision support intervention. (Stage III)

XIII. To evaluate patient-participants' perceived shared decision-making effort. (Stage III)

XIV. To evaluate the degree of decision support provided by provider-participants during an appointment with the patient-participant. (Stage III)

XV. To evaluate provider-participant assessments of both provider- and patient-directed decision support interventions. (Stage III)

XVI. To evaluate barriers, facilitators, and experiences of the patient-directed decision support intervention by conducting patient/caregiver-participant interviews. (Stage III)

XVII. To evaluate barriers, facilitators, and experiences of the provider-directed components intervention by conducting a focus group with providers. (Stage III)

XVIII. To evaluate the consent rate of patient-participants to germline testing. (Stage III)

OUTLINE:

OBSERVATIONAL STUDY (CLOSED TO ENROLLMENT)

STAGE I: San Francisco Veterans Affairs Health Care System (SFVAHCS) patients and providers participate in an audio recorded discussion on study. Patients also complete surveys and participate in interviews on study. Caregivers and providers also participate in interviews on study. Participants medical records are reviewed throughout the study.

STAGE II: Subset of SFVAHCS patients, caregivers, and providers who participated in stage I participate in an interview and may be asked to participate with an advisory board on study. Non-SFVAHCS providers participate in an interview on study.

INTERVENTIONAL STUDY:

STAGE III: About 14 days prior to scheduled germline testing appointment, patients and caregivers call or meet with a coach to select decision aid genetics adviser (GA) platform preference delivery (online, print, or both online and print), review the GA online platform, and possibly undergo consultation and training for audio recording of the scheduled appointment. Patients and caregivers attend the scheduled germline testing appointment on day 1. Patients complete surveys and patients and caregivers may complete an interview on study for up to 90 days post-appointment. Providers participate in focus groups and complete surveys on study and for up to 24 months.

ELIGIBILITY:
Stage 1: Inclusion Criteria

Patient-participants:

1. Age 18 years or older.
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Able to understand a written informed consent document and willing to sign it.
4. Able to speak, read, and understand English.
5. Documentation of locally advanced (pelvic lymph node-positive), metastatic, or castration-resistant prostate cancer in a clinical progress note or pathology report.
6. Scheduled to attend a hematology/oncology appointment (in person or remote) during which provider anticipates discussing germline testing, somatic tumor testing, or targeted therapy.

Caregiver-participants:

1. Age 18 years or older.
2. Identified by a patient-participant as an individual who is involved with the patient's care, and willing to join the interviews.
3. Able to provide verbal consent.
4. Able to speak and understand English.

Provider-participants:

1. Hematology/oncology or Genetics provider (medical doctor (MD) or nurse practitioner (NP), post-first year clinical fellows allowed).
2. Has discussed germline testing, somatic testing, or targeted therapy for an San Francisco Veteran Health Care System (SFVAHCS) patient with locally advanced or metastatic prostate cancer (as defined above) within the past 90 days of being contacted about the study.
3. Able to provide consent via email.

Stage 2: Inclusion Criteria:

Patient participants:

1. Participated in Stage 1.
2. Completed either germline or tumor testing for prostate cancer.
3. Able to understand study procedures and to comply with them for the entire length of the study.

Caregiver-participants:

1. Participated in Stage 1.
2. Partner, family-member, or friend of a Stage 2 participant (identified by the patient-participant as a caregiver).

SFVAHCS Provider-participants:

1. Participated in Stage 1.
2. Meets one of the two following criteria:

   * Physician specializing in medical oncology (MD, post-first year clinical fellows allowed) who has discussed genetic testing or targeted therapy with a patient with advanced prostate cancer within the past 30 days of being contacted for this study.
   * Physician specializing in genetics who has discussed genetic testing or targeted therapy with a patient with advanced prostate cancer within the past 90 days of being contacted for this study.

Non-SFVAHCS provider-participants:

1. Meets one of the three following criteria:

   * Principal investigator of a Precision Oncology Program for Cancer of the Prostate (POPCaP) site.
   * Physician specializing in medical oncology who has discussed genetic testing or targeted therapy with a patient with advanced prostate cancer within the past 30 days of being contacted for this study.
   * Physician specializing in genetics who has discussed genetic testing or targeted therapy with a patient with advanced prostate cancer within the past 90 days of being contacted for this study.

   Note: For Non-SFVAHCS providers, fellows are not eligible.
2. Able to understand study procedures and to comply with them for the entire length of the study.

Stage 3: Inclusion Criteria

Patient-participants

1. Age 18 years or older.
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Able to understand a written informed consent document and willing to sign it.
4. Able to speak, read, and understand English.
5. Documentation of high-risk localized, very high-risk localized, locally advanced (pelvic lymph node-positive), metastatic, or castration-resistant prostate cancer in a clinical progress note or pathology report.
6. Scheduled to attend a hematology/oncology appointment (in person or remote) during which provider anticipates discussing germline testing.

Caregiver-participants

1. Age 18 years or older.
2. Identified by a patient-participant as an individual who is involved with the patient's care, and willing to join the interview.
3. Able to provide verbal consent.
4. Able to speak and understand English.

Provider-participants

1. SFVAHCS physician (MD) trained in medical oncology or undergoing training as a clinical fellow.
2. Has discussed germline testing for prostate cancer with an SFVAHCS patient within the past year of being contacted about the study, or plans to discuss germline testing for prostate cancer with an SFVAHCS patient.
3. Able to provide verbal consent.

Stage 1: Exclusion Criteria

Patient-participants:

1. For patient-participants undergoing genetic testing, if results of the genetic tests have already been disclosed to the participant, they are not eligible.

   Caregiver and Provider-Participants
2. If they do not meet any of the inclusion criteria above.

Stage 2: Exclusion Criteria

1. Participants who do not meet the inclusion criteria above.

Stage 3: Exclusion Criteria

Patient-participants:

1. Prior receipt of germline testing.
2. Prior participation in Stage 1 for germline testing.

Caregiver and Provider-Participants

1. If they do not meet any of the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean score on the Decisional Conflict Scale (DCS) (Stage 1) | 6 months
  The Decisional Conflict Scale measures personal perceptions of : a) uncertainty in choosing options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. Scoring and interpretation Items are given a score value ranging from 0 = 'strongly disagree' to 4 = 'strongly agree'. Total Scores are a sum of the scores of the 16 items and are scaled by divided by 16 and then multiplied by 25 for a total scale score range from 0 [extremely high decisional conflict] to 100 [no decisional conflict]. Mean score and 95% confidence interval (CI) of the total DCS as well as the 4 subscales will be calculated.
Proportion of participants with a total score of >37.5 on the DCS (Stage 1) | 6 months
  Participants who completed the DCS will be divided by their total score into those who scored >37.5 or not. The proportion of participants with a total score of > 37.5 will be reported.
Proportion of participants enrolled (Stage 3) | Up to 3 years
  The proportion of invited participants who consent to the study compared to the total number of participants approached will be reported as measured by study entry.
Proportion of participants providing reason for not enrolling (Stage 3) | Up to 3 years
  The proportion of invited participants who do not consent to the study will have the reason for not joining recorded and totaled.

SECONDARY OUTCOMES:
Mean score on the germline testing knowledge scale (Stage 1) | 6 months
  Proportion of participants with correct responses on where participants response with an agree or disagree to each item addressing information they have received regarding germline testing. The proportion of participants who correctly responded to each knowledge item receive a score of 1 for a total score range of 0 - 16. Mean score and 95% CI of the total knowledge scale will be reported.
Mean change in germline testing knowledge score (Stage 3) | Up to 6 months
  The mean change in germline testing knowledge score from baseline to 7 days post appointment will be reported for participants in Stage 3. Participants with correct responses on where participants response with an agree or disagree to each item addressing information they have received regarding germline testing. The correct response to each knowledge item receives a score of 1 for a total score range of 0 - 16. Mean change in score and 95% CI of the total knowledge scale will be reported.
Proportion of participants with correct responses on germline testing knowledge scale | 6 months
  The germline testing knowledge scale is a 16 item survey where participants response with an agree or disagree to each item addressing information they have received regarding germline testing. The proportion of participants who correctly responded to each knowledge item and 95% CI for each knowledge item will be reported.
Mean score on the somatic testing knowledge scale | 6 months
  The somatic testing knowledge scale is a 17-item survey where participants response with an True, false, or don't know to each item addressing information they have received regarding personalized cancer therapy and molecular testing (target therapy). The proportion of participants who correctly responded to each knowledge item receive a score of 1 for a total score range of 0 - 17. Mean score and 95% CI of the total knowledge scale will be reported.
Proportion of participants with correct responses on the somatic testing knowledge scale | 6 months
  The somatic testing knowledge scale is a 16-item survey where participants response with an True, false, or don't know to each item addressing information they have received regarding personalized cancer therapy and molecular testing (target therapy). The proportion of participants who correctly responded to each knowledge item will be reported with 95%confidence intervals.
Proportion of patients for whom there was 'gold standard' shared decision making (collaboRATE) | 6 months
  The collaboRATE scale is a 3 item scale with responses ranging from 0 -10 for each item which ask the participant to think about the appointment they just had. These responses will be scored using the Top Score approach which excludes cases where a response to one or more of the collaboRATE questions is missing. Each encounter is coded as either '1', if the response to all three collaboRATE items was 9, or '0' if the response to any of the three collaboRATE items was less than 9. The percentage of all encounters that were coded as '1' is the collaboRATE Score. Higher scores represent more shared decision making. This number also corresponds to the proportion of patients for whom there was 'gold standard' shared decision making. Percentage and 95% CI will be calculated.
Mean Brief Decision Support Analysis Tool (DSAT-10) scores | 6 months
  The Brief Decision Support Analysis Tool (DSAT-10) will be used to evaluate treating physicians' and practitioners' use of decision support and communication skills for recordings (Guimond, et al. Patient Education Counsel 2003). Encounters are reviewed and scored on 5 factors such as Decision making status, Knowledge of, Values/Preference associated with, Others' involvement with the decision, and Next Steps and given a score ranging from 1-10, with a higher score indicating a greater quality of decisional support.The DSAT-10 will be applied to calculate a mean and 95% CI of the total score (0-10) and of the 5 factors.
Proportion of providers who responded to yes for pre-test germline testing items | 6 months
  In addition,to the regular germline testing questionnaire, the following provider communication items will be scored as Yes or No, based on 1.2022 National Comprehensive Cancer Network (NCCN) guidelines for pre-test germline testing: Prepare patient for possible outcomes of testing, including positive, negative, and variant of uncertain significance (VUS), Discuss possible management options if a mutation is identified, Advise about possible inherited cancer risk to relatives. Discuss cost of testing, Provide overview of current legislation regarding genetic, discrimination, Provide overview of current legislation regarding privacy of genetic, information, Discuss plan for results disclosure. Proportion of providers who responded yes to each item will be reported.
Proportion of providers who responded to yes for pre-test tumor testing item | 6 months
  In addition,to the regular germline testing questionnaire, the following provider communication item will be scored as Yes or No, based on 1.2022 NCCN guidelines for pre-test tumor testing: Prepare patient for possible outcomes of testing. Proportion of providers who responded yes will be reported.
Proportion of participants who received the precision oncology intervention or testing | 6 months
  The proportion of participants who received the precision oncology intervention or testing discussed during appointment as well as the type of intervention (germline, somatic, or targeted therapy) will be reported.
Mean change in score on the Decisional Conflict Scale (DCS) (Stage 3) | Up to 6 months
  The Decisional Conflict Scale measures personal perceptions of : a) uncertainty in choosing options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. Scoring and interpretation Items are given a score value ranging from 0 = 'strongly disagree' to 4 = 'strongly agree'. Total Scores are a sum of the scores of the 16 items and are scaled by divided by 16 and then multiplied by 25 for a total scale score range from 0 [extremely high decisional conflict] to 100 [no decisional conflict]. Mean score change and 95% confidence interval (CI) of the total DCS as well as the 4 subscales will be calculated between baseline and 7 days post appointment.
Proportion of research staff and providers who agree to participate (Stage 3) | Up to 6 months
  Adoption will be measured by the proportion of research staff and providers who agree to participate in the patient-directed decision support intervention divided by the number of invited providers.
Proportion of research staff who completed all components of the decision support intervention (Stage 3) | Up to 6 months
  The proportions of research staff who complete each component of the patient-directed decision support intervention for each eligible patient-participant:1) decision aid platform preference assessment; 2) decision aid delivery; 3) question list coaching; 4) summary and question routing; and 5) reminder message sending, measured by verbal questionnaire.
Proportion of providers who completed all components of the decision support intervention (Stage 3) | Up to 6 months
  The proportions of providers who complete each component of the provider-directed decision support intervention for each patient-participant: 1) teach back; 2) review and/or solicit questions; 3) discuss benefits of germline testing; and 4) discuss risks of germline testing, measured by analyzing the consultation audio recording.
Proportion of patient-participants who completely review the decision aid (Stage 3) | Up to 6 months
  The proportion of patient-participants who completely review the decision aid, measured by user analytics 7 days post-appointment will be reported.
Proportion of patient-participants who request training for audio-recording (Stage 3) | Up to 6 months
  The proportion of patient-participants who request training to audio-record their appointment who then create an audio recording, measured by questionnaire 7 days post-appointment will be reported.
Proportion of patient-participants who request question list coaching (Stage 3) | Up to 6 months
  The proportion of all patient-participants who request question list coaching and who then ask at least one question from the question list during their appointment, as measured by analyzing the consultation audio recording will be reported.
Proportion of participants with responses of 9-10 on the Net Promoter Score scale (Stage 3) | Up to 6 months
  The Net Promoter Score is a single item measure used to gauge satisfaction, and enthusiasm for the intervention. Total response options range from 0-10, with participants who select a response of 9 or 10 to be considered 'promoters". Responses will be obtained by questionnaire, 7 days post-appointment and the proportion of participants who respond with a choice of 9 or 10 will be reported.
Proportion of patient-participants who report "somewhat" or "very helpful" on evaluation of patient-directed intervention (Stage 3) | Up to 6 months
  The proportion of patient-participants who report "somewhat helpful" or "very helpful" in their evaluation of the patient-directed intervention, and each of its components, on 5-point Likert scale with responses options of "not helpful at all", "somewhat not helpful", "neither helpful nor not helpful", "somewhat helpful", and "very helpful" measured by questionnaire. 7 days post-appointment will be reported.
Proportion of provider-participants who report "somewhat agree" or "strongly agree" to any one of the components of the intervention (Stage 3) | Up to 6 months
  The proportion of provider-participants who report "somewhat" or "strongly agree" with the acceptability, feasibility, compatibility, simplicity, and relative advantage of the interventions, on a 5-point Likert scale with responses options of "strongly disagree", "somewhat disagree", "neither agree or disagree", "somewhat agree", and "strongly agree" measured by questionnaire.
Proportion of patient-participants who consent to germline testing (Stage 3) | Up to 3 years
  Proportion of patient-participants who consent to germline testing, by medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kwon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No